CLINICAL TRIAL: NCT02151604
Title: A Study to Determine Regional Lung Function in Patients With Non-small Cell Lung Cancer (NSCLC) Undergoing Radiotherapy Using Hyperpolarized Xenon Gas MR Imaging
Brief Title: Hyperpolarized Xenon Gas MR Imaging in NSCLC Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HPX-2011-003; 2011-002028-41 (EudraCT Number)
Record Dates: First submitted 2014-05-21; First posted 2014-05-30 (Estimated); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- 129 Xenon MR Imaging (Experimental): Xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Interventions: Drug: Inhalation of hyperpolarized xenon gas

INTERVENTIONS:
Drug: Inhalation of hyperpolarized xenon gas — The xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.

SUMMARY:
Lung cancer is the second most commonly diagnosed cancer in the United Kingdom, accounting for 22% of cancer deaths. The main treatments for lung cancer are surgery, radiotherapy or chemoradiotherapy. Current methods, for assessing lung function in lung cancer patients i.e. spirometry and gas transfer are inadequate. We aim to develop a new technique capable of describing regional lung abnormality using hyperpolarized xenon gas MRI.

The study will involve 50 patients diagnosed with lung cancer considered suitable for radical radiotherapy or chemoradiotherapy. Participants will be offered hyperpolarized Xe129 MR at baseline, two weeks after commencement of radiotherapy schedules and four followup visits over one year posttreatment.

Patients will undertake extensive study measures at baseline and followup visits, including chest CT scans, ventilation/perfusion nuclear medicine scans, gadolinium enhanced MRI scans, pulmonary function tests, breathlessness scores, radiotherapy induced lung toxicity assessments and exercise testing. Participation in these full tests takes a day, allowing patients time to rest between tests and allowing for a period of observation following the final hyperpolarized xenon scan.

The investigators will correlate baseline hyperpolarized Xe129 MR imaging with spirometry and breathlessness scores to determine if tolerance for radiotherapy is better predicted by hyperpolarized Xe129 MR imaging. The investigators will evaluate changes in hyperpolarized Xe129 MR imaging before and after radiotherapy (RT) to determine if it provides better monitoring of response compared with spirometry.

The study will take place at the Churchill Hospital, Oxford University Hospitals National Health Service Trust and will be funded by the National Institute for Health Research Oxford Biomedical Research Centre. Hyperpolarized Xe129 MR imaging has the potential to inform individual suitability for radiotherapy schedules better than the investigations used currently. In addition, hyperpolarized Xe129 MR imaging has the potential for better monitoring of treatment response and improved detection of radiation induced lung injury, invaluable to treating patients with radiation induced injury.

DETAILED DESCRIPTION:
Survival rates for lung cancer are poor. One year survival rate in the United Kingdon for males is 27% and for females 30%, falling to less than 10% at five years. Prognosis for lung cancer is so poor because over two thirds of patients are diagnosed at a late stage when curative treatment is not possible. Early diagnosis and assessment of tolerance for curative treatment would make a significant difference to survival rates.

Histologically, approximately 80% of lung cancer is nonsmall cell lung cancer (NSCLC). The main curative treatment for NSCLC is surgery. Radical radiotherapy and chemoradiotherapy are other potentially curative treatments. These are suitable for patients who present with localized tumours that are surgically unresectable due to involvement of critical local structures or medically inoperable disease due to advanced age or comorbidities. Radiotherapy aims to deliver a high tumouricidal dose to the tumour without damaging the surrounding normal lung tissue. A high dose of radiotherapy improves local control but incurs a risk of inducing toxic effects in the normal lung tissue. If radiationinduced lung toxicity could be better predicted and monitored, radical radiotherapy could be tailored to the individual, which could also have the benefit of avoiding or reducing radiation dose to functional lung tissue.

Currently assessment of patients for radiotherapy involves lung function measurements to provide a clinical indicator as to whether or not the patient would tolerate treatment and maintain sufficient functioning lung posttreatment to continue with activities of daily living without significant impairment. The current gold standard for assessment of lung function is spirometry and gas transfer. Spirometry and gas transfer measure global lung function but provides no information about the different regions of the lung or regarding the support 'framework' of the lung, the parenchyma.Changes in lung function as measured by spirometry or gas transfer do not coherently correlate with symptom severity or reflect a decline in patient health. This weak relationship is probably because the lung is a complex regional organ where localized disturbances of a variety of factors including gas flow (ventilation), blood flow (perfusion) and gas transfer all combine to impair respiratory function.

To address these issues we aim to use hyperpolarized xenon gas (Xe129) magnetic resonance imaging (MRI)and computed tomography (CT)to describe detailed regional and structural lung abnormality in patients with NSCLC. The investigators will correlate this technique with baseline spirometry and dyspnoea scores to determine if respiratory tolerance of radiotherapy is better predicted by hyperpolarized Xe129 MR imaging. The investigators will compare hyperpolarized Xe129 MRI with standard imaging(nuclear medicine scans). The investigators will also evaluate changes in hyperpolarized Xe129 MR imaging before, during and after radiotherapy to determine if it provides improved assessment of radiationinduced lung injury. MRI has advantage of being free from ionizing radiation making it safe and practical for diseases like lung cancer where repeated followup scans are necessary. MR imaging has an enhanced speed of image acquisition compared with CT and lung scintigraphy and offers the potential of dynamic assessment of lungs during respiration. In conventional MRI, the signal originates principally from the protons in water molecules of tissues. Therefore conventional MRI has limited use in respiratory disease because the lung has a very low density of protons, instead being largely composed of air spaces that do not generate MR signal. Hyperpolarised noble gases can resolve this problem. Xenon (Xe129) is an unreactive or inert noble gas. It has a nuclear spin of ½ enabling use in MR imaging to generate a signal. Xe129 is hyperpolarized, that is to say that nuclear spin within the atoms is increased. Hyperpolarization increases the MR signal enabling the Xe129 gas to show up on the MR scan. In portions of the lung that have good airflow, the hyperpolarized Xe129 gas will show up more and be seen more quickly. In addition Xe129 readily dissolves in blood where it emits different MR signal characteristics. This property may be exploited to regionally quantify both ventilation and perfusion within the lung providing a comprehensive assessment of lung function. The need for improved functional imaging to identify preexisting lung disease and predict respiratory tolerance of patients with NSCLC for radiotherapy treatment is clear. Hyperpolarized Xe129 MR imaging has the potential to inform individual suitability for radiotherapy schedules better than the investigations used currently. In addition improved functional imaging is required to monitor treatment response and enable treatment regimes to be tailored to the individual. Hyperpolarized Xe129 MR imaging offers the potential of improved detection of radiationinduced lung injury, invaluable to treating patients with radiation induced injury. It may also provide information that would allow RT to be planned in such a way as to reduce the risk of patients developing radiationinduced lung toxicity (RILT).

The need for improved functional imaging to identify preexisting lung disease and predict respiratory tolerance of patients with NSCLC for radiotherapy treatment is clear. Hyperpolarized Xe129 MR imaging has the potential to inform individual suitability for radiotherapy schedules better than the investigations used currently. In addition improved functional imaging is required to monitor treatment response and enable treatment regimes to be tailored to the individual. Hyperpolarized Xe129 MR imaging offers the potential of improved detection of radiationinduced lung injury, invaluable to treating patients with radiation induced injury. It may also provide information that would allow RT to be planned in such a way as to reduce the risk of patients developing radiationinduced lung toxicity (RILT).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or Female, aged 18 years or above
* Histologically verified NSCLC
* Patients with any stage NSCLC where radical radiotherapy (with either conventionally fractionated treatment or with stereotactic body radiotherapy (SABR)) or chemoradiotherapy (concurrent or sequential schedule) is considered appropriate
* WHO performance status 0-2
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Inability to give written informed consent
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Previous radiotherapy to the chest
* The presence of another condition where the disease itself or treatment may interfere with the study endpoints
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Inability to lie flat for imaging
* Contraindications to MRI examination including indwelling pacemaker, non-MRI compatible metallic implant, severe claustrophobia, intra-ocular foreign body
* Contraindications for gadolinium enhanced lung MRI scan - known hypersensitivity/allergy to the injection of MultiHance (contains gadobenate dimeglumine and small quantities of benzyl alcohol) that is given as part of this scanning or an adverse reaction to an injection given during previous MRI scanning, severe renal impairment
* Contraindications for ventilation/perfusion nuclear medicine scanning - known hypersensitivity to albumin or preference to avoid blood donation product
* Epilepsy requiring on-going medical treatment, or a seizure within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fergus V Gleeson, MB BS, FRCP, Principal Investigator — Professor of Radiology
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the lung cancer oncology clinics by the oncology team Recruitment period: 23/04/2014 to 30/11/2019
Pre-assignment Details: All participants were recruited to one arm. No control or comparative cohort in this study
Groups:
- 129 Xenon MR Imaging Group: Xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Inhalation of hyperpolarized xenon gas: The xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Patients with cancer with planned radiotherapy to their thorax which may affect their lungs.
  Up to 6 xenon scans per visit at baseline (pre-treatment), mid-point, end of radiotherapy and 4 weeks after. Patientswith lung cancer would already receive CT chest at the baseline, end-of-treatment visits and 4 weeks after that.
Period: Overall Study
Arm/Group | 129 Xenon MR Imaging Group
Started | 22
Completed | 13
Not Completed | 9
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Not all participants have had their baseline measurements taken due to a number of interim ethics approved study amendments and some logistic issues. But age, sex, CT and HPXMRI were acquired for all patients enrolled in the study.
Arm/Group | 129 Xenon MR Imaging
Number analyzed (Participants) | 22
Age, Continuous [Median (Standard Deviation); unit: years] | 72.10 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 22
Pulmonary Function Tests [Count of Participants; unit: Participants] | 11
Ventilation/perfusion nuclear medicine scan (optional) [Count of Participants; unit: Participants] | 0
Computed Tomography (CT) of the Chest [Count of Participants; unit: Participants] | 14
Hyperpolarized Xe-129 MR Imaging [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change From Baseline in Ventilation Map Using Hyperpolarized Xe-129 MR Imaging
Description: Number of participants with a change from baseline in ventilation map using hyperpolarized Xe-129
Time Frame: Mid-point of radiotherapy - varies depending on the duration of treatment prescribed, between 1 week to 2 months from the baseline scan (range: 7 days to 60 days). For example, for 2 weeks of radiotherapy, this would be at 1 week post-baseline.
Population: 10 patients had at least one follow-up after baseline
Measure: Count of Participants; unit: Participants
Groups:
- 129 Xenon MR Imaging Group: Xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Inhalation of hyperpolarized xenon gas: The xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Patients with cancer with planned radiotherapy to their thorax which may affect their lungs.
  Up to 6 xenon scans per visit at baseline (pre-treatment), mid-point, end fo radiotherapy and 4 weeks later.
  Lungg cancer patients would already receive CT chest at the baseline and end-of-treatment visits and 4 weeks follow-up.
Arm/Group | 129 Xenon MR Imaging Group
Number analyzed (Participants) | 10
Participants | 6
Statistical Analysis 1: Comparison: 129 Xenon MR Imaging Group; Correlation with field of irradiation; Test type: Other; p = 0.041, Pearson's correlation analysis; Pearson's coefficient = -0.57

2. Secondary Outcome: Number of Participants With a Change in Ventilation and ADC Maps Using Hyperpolarized Xe-129 MR Imaging From Baseline to 3 Months Post Radiotherapy Completion
Description: Number of participants with a change in ventilation MRI acquired for 5 patients, 3 months after treatment completion ADC not acquired in this study
Time Frame: 3 months after completion of treatment
Population: Ventilation MRI acquired for 5 patients 3 months after treatment completion
Measure: Count of Participants; unit: Participants
Groups:
- 129 Xenon MR Imaging Group: Xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Inhalation of hyperpolarized xenon gas: The xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Patients with cancer with planned radiotherapy to their thorax which may affect their lungs.
  Up to 6 xenon scans per visit at baseline (pre-treatment), mid-point, end of radiotherapy and 3 months after. Patientswith lung cancer would already receive CT chest at the baseline, end-of-treatment visits and 3 months after that.
Arm/Group | 129 Xenon MR Imaging Group
Number analyzed (Participants) | 5
Participants | 3

3. Secondary Outcome: Correlation Between Change in Ventilation/ ADC Maps Using Hyperpolarized Xe-129 MR Imaging and Change in Lung Function From Baseline to Follow-up (During Treatment)
Description: Correlation between change in ventilation or ADC maps using hyperpolarized Xe-129 MR imaging and change in lung function from baseline to follow-up (during treatment), acquired at the mid-point of treatment.
Time Frame: Mid-point of radiotherapy - varies depending on the duration of treatment prescribed, between 1 week to 2 months from the baseline scan - Range: 7-60 days.) For example, for 2 weeks of radiotherapy, this would be at 1 week post-baseline.
Population: Participants with mid-point follow-up
Measure: Number; unit: Pearson's Coorelation Coefficient
Arm/Group | 129 Xenon MR Imaging Group
Number analyzed (Participants) | 10
Pearson's Coorelation Coefficient
  Alveolar volume (VA) | 0.60
  Diffusing capacity for carbon monoxide(TLCO) | 0.70
  Residual volume (RV) | -0.85
  Functional residual capacity (FRC) | -0.95
  Inspiratory capacity(IC) | -0.88
Statistical Analysis 1: Comparison: 129 Xenon MR Imaging Group; Correlation of change in ventilation signal with that of alveolar volume (VA); Test type: Other; p = 0.037, Pearson's Correlation Analysis — Pearson's correlation coefficient: 0.60; 0.60; Pearson's coefficient = 0.60
Statistical Analysis 2: Comparison: 129 Xenon MR Imaging Group; Correlation of change in ventilation signal with that of diffusing capacity for carbon monoxide(TLCO); Test type: Other; p = 0.012, Pearson's correlation analysis; Pearson's correlation coefficient: 0.70; Pearson's correlation coefficient = 0.70
Statistical Analysis 3: Comparison: 129 Xenon MR Imaging Group; Correlation of change in ventilation signal with that of residual volume (RV); Test type: Other; p = 0.032, Pearson's correlation analysis; R = -0.85; Pearson's correlation coefficient = -0.85
Statistical Analysis 4: Comparison: 129 Xenon MR Imaging Group; Correlation of change in ventilation signal with that of functional residual capacity (FRC); Test type: Other; p = 0.004, Pearson's correlation analysis; R = -0.95; Pearson's correlation coefficient = -0.95
Statistical Analysis 5: Comparison: 129 Xenon MR Imaging Group; Correlation of change in ventilation signal with that of inspiratory capacity(IC); Test type: Other; p = 0.012, Pearson's correlation analysis; Pearson's correlation coefficient = -0.88; Pearson's correlation coefficient = -0.88

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the participants from the time of the first bag of xenon inhaled until 2 weeks after the date of the last scan, up to 6 months
Description: Standard definitions apply.
  All AEs observed by the investigator or reported by the patient during and for 24 hours following xenon MRI are reported. Only adverse events where there is a reasonable possibility of a relationship to xenon, and any adverse event considered to be of medical interest/ importance are reported. Description, date of onset and end date, severity, assessment of relatedness to trial medication, other suspect drug or device and action taken will be recorded.
Groups:
- 129 Xenon MR Imaging Group: Xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Inhalation of hyperpolarized xenon gas: The xenon gas is inhaled immediately before acquisition of an MR image to enable the lung structure to be seen.
  Patients with cancer with planned radiotherapy to their thorax which may affect their lungs.
  Up to 6 xenon scans per visit at baseline (pre-treatment), mid-point, and end fo radiotherapy. Patients would already receive CT chest at the baseline and end-of-treatment visits.
Arm/Group | 129 Xenon MR Imaging Group
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 14/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 129 Xenon MR Imaging Group (N=22)
Dizziness (Nervous system disorders) | 8 (19)
Dysgeusia (Nervous system disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Euphoria (Nervous system disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hypersalivation (Gastrointestinal disorders) | 1 (1)
Chest tightness (Reproductive system and breast disorders) | 1 (1)
Paresthesia (Lips) (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
3 patients were recruited prior a substantial amendment was put in place thus were excluded from the analysis due to different study objectives being in place at that time.

4 patients were not able to breath hold during the MRI scan and therefore good quality image scans of their lungs could not be obtained on those occasions. The scans were excluded from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02151604/Prot_SAP_000.pdf